CLINICAL TRIAL: NCT03748485
Title: Comparing the Treatment Efficacy in Clinical Local Advanced Colorectal Cancer (cTxN1/2M0) Following Preoperational Adjuvant Therapies and Pathologically Proved StageⅡ(pT0-3N0M0)With or Without Adjuvant Chemotherapy
Brief Title: Adjuvant Chemotherapy in Clinical Local Advanced CRC Following Preoperational Therapies and pT0-3N0M0 Diagnosis
Acronym: CANWATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianping Wang, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L2018ZSLYEC-162
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Adjuvant Chemotherapy
Keywords: local advanced colorectal cancer; adjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wait and watch group (Experimental): clinical local advanced colorectal cancer (cTxN1/2M0) following pre-operational adjuvant therapies and pathologically proved stageⅡ(pT0-3N0M0) without adjuvant chemotherapy
  Interventions: Behavioral: wait and watch
- adjuvant chemotherapy group (Active Comparator): clinical local advanced colorectal cancer (cTxN1/2M0) following preoperational adjuvant therapies and pathologically proved stageⅡ(pT0-3N0M0) with adjuvant chemotherapy
  Interventions: Drug: adjuvant chemotherapy

INTERVENTIONS:
Behavioral: wait and watch — clinical local advanced colorectal cancer (cTxN1/2M0) following preoperational adjuvant therapies and pathologically proved stageⅡ(pT0-3N0M0),without(wait and watch) adjuvant chemotherapy
  Arms: wait and watch group
Drug: adjuvant chemotherapy — clinical local advanced colorectal cancer (cTxN1/2M0) following preoperational adjuvant therapies and pathologically proved stageⅡ(pT0-3N0M0),with adjuvant chemotherapy
  Other Names: mFOLFOX6
  Arms: adjuvant chemotherapy group

SUMMARY:
Adjuvant chemotherapy was unnecessary in pathological stage Ⅱ colorectal cancer following initial treatment of surgery without high risk factors of recurrences. The treatment efficacy of adjuvant chemotherapy for pT1-3N0M0 colorectal cancer following preoperational chemotherapy or chemoradiotherapy remains unclear. Part of clinical local advanced colorectal cancer(cTxN1-2M0), which turn out to be pT0-3N0M0 after preoperational chemotherapy or chemoradiotherapy, might not really need adjuvant chemotherapy due to the down-stage efficacy of the preoperational treatments, or the misleading by lymph nodes false-positive imaging diagnosis.

DETAILED DESCRIPTION:
Colorectal cancer(CRC) nowadays rank the 3rd incidence and the 4th mortality in all cancers worldwide(ref). Although the coloscopy or liquid biopsy screen has improved the early diagnosis of CRC, about 26.5-36.0% of the patients were diagnosed local advanced CRC at the first visit. Part of clinical local advanced colorectal cancer(cTxN1-2M0), which turn out to be pT1-3N0M0 after preoperational chemotherapy or chemoradiotherapy, might not really need adjuvant chemotherapy due to the down-stage efficacy of the preoperational treatments, or the misleading by lymph nodes false-positive imaging diagnosis. Adjuvant chemotherapy was been admitted unnecessary in the pathological stage ⅡA (pT0-3N0M0) CRC following initial treatment of surgery without high risk factors of recurrences. The treatment efficacy of adjuvant chemotherapy for pT1-3N0M0 CRC following preoperational chemotherapy or chemoradiotherapy remains unclear. The aim of this study is to evaluate the efficacy/safety of adjuvant chemotherapy in clinical local advanced CRC (cTxN1/2M0) following preoperational adjuvant therapies and pathologically proved pT0-3N0M0 CRC. Patients are randomized to control group(down-staged pT0-3N0M0 CRC with 6 to 8 periods adjuvant chemotherapy) and experimental group(watch group, down-staged pT0-3N0M0 CRC without adjuvant chemotherapy). The primary endpoint is the 3-years disease-free survival after surgery. Secondary endpoints evaluate long-term clinical outcomes, in particular overall survival and side effect of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* preoperative clinical tumor stage III （TxN1-2M0）CRC
* pathological proved CRC adenocarcinoma by endoscopic biopsy
* Post operational pathological T0-3N0M0 without high risk factors of recurrence
* Patient able to understand and sign written informed consent

Exclusion Criteria:

* Other malignant tumors history.
* Complications need emergency surgery (occlusion, sub-occlusion, massive hemorrhage and abscesses).
* Colorectal tumor extension towards abdominal wall and/or adjacent organ making liver R0 resection impossible immediately.
* Non resectable lymph node metastasis.
* American Society of Anesthesiologists (ASA) grading≥ IV and/or, Eastern Cooperative Oncology Group(ECOG) score≥ 2.
* Physical or psychological dependence.
* Pregnant or breast feeding women.
* Not controlled pre-operational infection.
* Enrolled in other clinical trials within 4 weeks.
* Other clinical or laboratorial condition not recommended by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3years
  3years disease-free survival rate

SECONDARY OUTCOMES:
overall survival | 5years
  5years overall survival rate
adverse reaction of adjuvant therapies | 3years
  Rate of participants with myelosuppression, gastrointestinal reaction, infection, lose hair
remission rate of adjuvant therapies | 1year
  CRC remission evaluation using RECIST after adjuvant therapies
death rate within 30 days post surgery | 30days
  death related directly with operation within 30 days
complication in 30 days post surgery | 30days
  Rate of participants with complications such as bleeding，infection，anastomotic fistula,etc

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wang, MD/PHD, Study Chair — sixth affiliate hospital of Sun yatsen Hospital
Locations (1):
- Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No